CLINICAL TRIAL: NCT02097212
Title: Correlation Between Trachebroncho Malacia/Hyperdynamic Airway Collapse And Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS#-2794
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Trachebronchomalacia (TBM); Hyper Dynamic Airway Collapse (HDAC); Obstructive Sleep Apnea (OSA)
Keywords: Tracheobronchomalacia; TBM; HyperDynamic Airway Collapse; HDAC; Obstructive Sleep Apnea; OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tracheobronchomalacia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that there is a strong correlation between OSA and TBM/HDAC. Our hypothesis is based on the similarities in mechanism (airway collapse), symptoms (daytime and nocturnal dyspnea) predisposing conditions (obesity and neuromuscular abnormalities of the chest wall and the diaphragm), and effect of interventions (CPAP and BIPAP) in these diseases.

DETAILED DESCRIPTION:
Tracheobronchomalacia (TBM) and HyperDynamic Airway Collapse (HDAC) are two distinct airway diseases that lead to airway collapse which can in turn lead to the symptoms of dyspnea, cough, and inability to expectorate sputum effectively. TBM entails flaccid tracheal and bronchial cartilages leading to airway collapse, emanating primarily from the anterior wall of the lumen. It is seen in conditions such as Relapsing Polychondritis and saber sheath tracheal deformity. HDAC on the other hand is the hyper-flaccidity of the membranous portion of the tracheobronchial tree leading to airway collapse. This condition is commonly seen with obesity and severe emphysema. TBM and HDAC frequently coexist.

In patients with TBM/HDAC sleep disorders are common. Patients often complain of poor quality sleep, snoring, daytime fatigue, and somnolence. These patients are often diagnosed with Obstructive Sleep Apnea (OSA) upon workup.

ELIGIBILITY:
Inclusion Criteria:

* Females and males ages 18-80 years old
* Able and willing to provide written informed consent
* Existing diagnosis of TBM or HDAC or both
* No pre-existing diagnosis of OSA
* No history of reconstructive surgery of chest wall or diaphragm

Exclusion Criteria:

* Inability to provide informed consent
* Non-English speaking
* Poorly controlled congestive heart failure
* Untreated Insomnia
* Severe Coronary artery disease with active symptoms of angina
* Patient is pregnant, or plans to become pregnant in next 3 months
* Moderate to severe bronchiectasis
* Severe untreated gastroesophageal disease (GERD).
* Moderate to large hiatal hernia deemed to be atleast in part responsible for TBM/HDAC
* Airway obstruction not caused by TBM /HDAC or secondary TBM/HDAC caused by conditions such as Chronic Obstructive Pulmonary Disease (COPD).
* Active or recent (with in last one year) cancer or cancer therapy (chemotherapy, radiation therapy or surgery)
* Inability to properly perform the home sleep test
* Unreliable test data after 2 attempts
* BMI>45

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this pilot study we plan to recruit 30 consecutive patients with TBM/HDAC from the interventional pulmonology clinic at National Jewish Health (NJH). These patients will already have an established diagnosis of TBM and/or HDAC.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale | Baseline
  The Epworth Sleepiness Scale is widely used in the field of sleep medicine as a subjective measure of a patient's sleepiness. The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing.

CONTACTS AND LOCATIONS:
Overall Officials: Ali I Musani, MD, FCCP, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Murgu SD, Colt HG. Tracheobronchomalacia and excessive dynamic airway collapse. Respirology. 2006 Jul;11(4):388-406. doi: 10.1111/j.1440-1843.2006.00862.x. PMID 16771908
- [Background] Majid A, Fernandez L, Fernandez-Bussy S, Herth F, Ernst A. [Tracheobronchomalacia]. Arch Bronconeumol. 2010 Apr;46(4):196-202. doi: 10.1016/j.arbres.2009.10.011. Epub 2009 Dec 9. Spanish. PMID 20004507